CLINICAL TRIAL: NCT05892848
Title: Evaluation of Some Biochemical Markers of Bone Turnover in Childern and Adolescents With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hager Momen Ismail, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-23-05-03MS
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases group: childern and adolescents with type 1 diabetes
  Interventions: Diagnostic Test: serum ostecalcin,serum sclerostin and parathroid profile
- control group: age and sex matched control childern and adolsecents
  Interventions: Diagnostic Test: serum ostecalcin,serum sclerostin and parathroid profile

INTERVENTIONS:
Diagnostic Test: serum ostecalcin,serum sclerostin and parathroid profile — evaluation of bone turnover markers in blood

SUMMARY:
Type 1 diabetes is associated with many longterm complications as retinopathy,neuropathy and nephropathy. Recently, several studies have linked type 1 diabetes to bone fragility.Studies conducted on patients with type 1 diabetes have concluded that bone is negatively affected in type 1 diabetes with impaired bone density,increased fracture risk and impaired bone turnover markers.

ELIGIBILITY:
Inclusion Criteria:

* childern and adolsecents below 16 years of age diagnsed with type 1 diabetes for at least 1 year age and sex-matched control childern and adolsecents will be included

Exclusion Criteria:

* childern and adolescents with congenital bone disease, those with disorders of the parathyroid gland and those with chronic kidney disease.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: childern and adolsecents below 16 years of age diagnsed with type 1 diabetes for at least 1 year age and sex-matched control childern and adolsecents will be included
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-10 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
level of serum ostecalcin, sclerostin in patients with type 1 diabetes ann d their age and sex matched control | 12 months
  markers of bone turnover in patients with type 1 diabetes and their matched control

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Starup-Linde J, Hygum K, Harslof T, Langdahl B. Type 1 Diabetes and Bone Fragility: Links and Risks. Diabetes Metab Syndr Obes. 2019 Dec 3;12:2539-2547. doi: 10.2147/DMSO.S191091. eCollection 2019. PMID 31819579
- [Background] Madsen JOB, Herskin CW, Zerahn B, Jensen AK, Jorgensen NR, Olsen BS, Svensson J, Pociot F, Johannesen J. Bone turnover markers during the remission phase in children and adolescents with type 1 diabetes. Pediatr Diabetes. 2020 Mar;21(2):366-376. doi: 10.1111/pedi.12963. Epub 2019 Dec 27. PMID 31840392
- [Background] El Amrousy D, El-Afify D, Shabana A. Relationship between bone turnover markers and oxidative stress in children with type 1 diabetes mellitus. Pediatr Res. 2021 Mar;89(4):878-881. doi: 10.1038/s41390-020-01197-5. Epub 2020 Oct 10. PMID 33038875
- [Background] Roh JG, Yoon JS, Park KJ, Lim JS, Lee HS, Hwang JS. Evaluation of bone mineral status in prepuberal children with newly diagnosed type 1 diabetes. Ann Pediatr Endocrinol Metab. 2018 Sep;23(3):136-140. doi: 10.6065/apem.2018.23.3.136. Epub 2018 Sep 28. PMID 30286569